CLINICAL TRIAL: NCT06548165
Title: Physiological Reaction After Food Intake
Acronym: NutriPulse
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Martin Heni, Prof. Dr. med. Martin Heni, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 168/24
Record Dates: First submitted 2024-08-06; First posted 2024-08-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Physiological Reactivity to Cues
Keywords: wearables; food intake; physiologic reaction
MeSH Terms: interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearables (Experimental): Participants will wear at least three sensors for the measurement of different physiological outcomes (heat rate variability, skin conductance, pulserate) for two weeks. Women can use a fourth sensor to measure the body core temperature intravaginally. Food intake will be assessed via photos.
  Interventions: Device: Wearable

INTERVENTIONS:
Device: Wearable — Participants will wear an electrode on the chest for the measurement of the heart rate variability, a sensor for temperature measurement, and a sensor for continuous blood glucose measurement. Food intake will be recorded via pictures. One mixed meal tolerance test will be performed as a reference for further analyses. Females have the option to use a device for intravaginal temperature measurement.

SUMMARY:
The goal of this clinical trial is to clarify the normal response of the body after food intake.

Therefore, participants will wear three wearables for two weeks and document their food intake via an app- and picture-based protocol.

DETAILED DESCRIPTION:
The aim of this study is to investigate physiologically measurable reactions of the body to food intake. We want to find out which of the parameters collected can provide information about food intake and which techniques for data collection are expedient in this context. Ultimately, the aim is to develop a way of determining food intake from physiological data from physiological data without the user indicating this to the device.

The following data is collected continuously over a period of 2 weeks: Electrocardiogram (ECG), pulse rate from photoplethysmogram, body temperature, movement, skin conductance, and a continuous glucose measurement in the interstitium (CGM). The test subjects will also be asked to document each of their meals and snacks via an app using a photo. As an optional additional examination, female study participants will be offered an intravaginal temperature measurement. This independently performed measurement enables the core body temperature to be recorded.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 25 kg/m2

Exclusion Criteria:

* vegan diet
* any kind of special diet, e.g. to lose weight
* use of medication, except for thyroid hormones and contraceptives

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Electrocardiogram | 2 weeks
  Changes in heart rate variability in response to food intake. Assessed through Vivalink ECG wearable that measures a continuous 3-channel ECG.
Body temperature | 2 weeks
  Changes in body temperature in response to food intake. Vivalink ECG and CORE sensor continuously measure the skin temperature. CORE sensor is also able to determine the body core temperature via a heat flux sensor. For women, body core temperature can be measured with the trackle wearable.
Skin conductance | 2 weeks
  Changes in skin conductance in response to food intake. CardioWatch wearable continuously measures the skin conductance
Glucose level | 2 weeks
  Changes in glucose levels in the interstitium in response to food intake. FreeStyle libre sensors continuously measure the glucose levels.

SECONDARY OUTCOMES:
Physical Activity | 2 weeks
  The wearable Vivalink ECG contains an accelerometer to continuously assess activity, intensity and body position.
Food intake | 2 weeks
  Assessed through photo-documentation of consumed food

OTHER OUTCOMES:
Correlation of physiological measures (electrocardiogram, pulserate, body temperature, skin conductance, glucose level) | 2 weeks
  Correlation of the obtained physiological measures (electrocardiogram, pulserate, body temperature, skin conductance, glucose level) among each other and with food quantity and quality will be assessed
Sex differences | 2 weeks
  Differences in the obtained physiological measures between sexes will be analyzed.
Correlation with glycemic and insulin sensitivity | 2 weeks
  Correlation of the obtained physiological measures among with glycemic, lipidemia, and insulin sensitivity will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heni, MD, Principal Investigator — University of Ulm
Locations (1):
- Universityhospital Ulm, Ulm, Germany